CLINICAL TRIAL: NCT05998954
Title: QLESP Block for Postoperative Analgesia in Hip Surgery
Brief Title: QLESP Block in Hip Surgery
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No patients enrolled
Sponsor: Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Xi Wu, Doctor, Huazhong University of Science and Technology
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: XH20230812
Record Dates: First submitted 2023-08-13; First posted 2023-08-21 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Dental Occlusion

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Transmuscular quadratus lumborum and modified erector spinae plane (QLESP) block (QLESP group) (Experimental): The patient was turned to the lateral decubitus position with the side to be blocked upward and a low-frequency curved array transducer was placed on the ﬂank cranially to the iliac crest to identify the transverse process of L4, quadratus lumborum muscle, erector spinae muscle, and psoas muscle. The needle was advanced to gently contact the transverse process using an in-plane technique and 15 ml of 0.375% ropivacaine was administered between the erector spinae muscle and the transverse process. The needle was subsequently withdrawn and redirected toward the interfascial plane between the quadratus lumborum and the psoas major muscles, where 15 ml of 0.375% ropivacaine was injected with repeated negative aspiration.
  Interventions: Procedure: transmuscular quadratus lumborum and modified erector spinae plane (QLESP) block
- Suprainguinal fascia iliaca block (SFI group) (Active Comparator): With the patient in the supine position, the ultrasound transducer was placed in a parasagittal orientation over the inguinal ligament, inferior medially to the anterior superior iliac spine. Using real-time ultrasound imaging internal oblique, sartorius and iliacus muscles, covered by the fascia iliacus, were identified. With the needle tip placed beneath the fascia and above the iliacus muscle from caudad-to-cephalad direction (in-plane technique), 30 ml of 0.375% ropivacaine was injected slowly to separate the fascia iliaca from the iliacus muscle.
  Interventions: Procedure: suprainguinal fascia iliaca block

INTERVENTIONS:
Procedure: transmuscular quadratus lumborum and modified erector spinae plane (QLESP) block — Fifteen ml of 0.375% ropivacaine was administered between the erector spinae muscle and the transverse process. Fifteen ml of 0.375% ropivacaine was subsequently given between the quadratus lumborum and the psoas major muscles.
  Arms: Transmuscular quadratus lumborum and modified erector spinae plane (QLESP) block (QLESP group)
Procedure: suprainguinal fascia iliaca block — Thirty ml of 0.375% ropivacaine will be injected cranial to the inguinal ligament between the fascia iliaca and the iliopsoas muscle.
  Arms: Suprainguinal fascia iliaca block (SFI group)

SUMMARY:
Total hip arthroplasty (THA) is a common surgical procedure aiming to improve mobility and quality of life in patients suffering from hip pain. Regional analgesia techniques are critical components of an optimal multimodal analgesia technique for THA, as they have been shown to improve pain relief as well as reduce opioid requirements. Ultrasound-guided suprainguinal fascia iliaca (SFI) block has been recommended as a reliable analgesic option for THA. However, SFI block may lead to decreased motor strength of the surgical limb thereby hindering postoperative mobilization. Recently, our group has developed a novel transmuscular quadratus lumborum and modified erector spinae plane (QLESP) block, which is characterized by simple operation, high efficiency, and wide dermatomal coverage of sensory block. In this randomized trial, we aimed to compare ultrasound-guided QLESP with SFI block as a component of non-opioid analgesic regimen in patients undergoing THA. The primary outcome of the study was postoperative sufentanil consumption within the initial 24-h postoperative period after THA. The secondary objectives were to compare pain scores, postoperative quadriceps strength, the time to first rescue analgesia, opioid-related adverse effects, time to ambulation, and the time to hospital discharge.

ELIGIBILITY:
Inclusion Criteria:

* 1. Age 18-65 yrs 2. American Society of Anesthesiologists classification 1-3 3. Body mass index between 20 and 35 (kg/m2) 4. Undergo elective primary unilateral THA via a posterolateral approach 5. Informed consent

Exclusion Criteria:

* 1. A known allergy to the drugs being used 2. Pre-existing neuropsychiatric disorders or language barrier 3. Analgesics intake, history of substance abuse 4. Contraindications to peripheral nerve block 5. Acute cerebrovascular disease 6. Severe liver failure

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-08-22 (Actual); Primary Completion 2024-08-20 (Estimated); Study Completion 2024-10-20 (Estimated)

PRIMARY OUTCOMES:
The cumulative opioid consumption | At 24 postoperative hours

SECONDARY OUTCOMES:
The pain scores determined by the numeric rating scale (NRS, 0-10) | At 1, 6, 12, 24, and 48 hours after the surgery
Quadriceps strength | At 1, 6, 12, 24, and 48 hours after the surgery
The time to first rescue analgesia | Within postoperative 48 hours
Postoperative hospital length of stay | Up to 6 weeks
The Time to Ambulation | Postoperative 48 hours
Adverse events | Postoperative 48 hours

CONTACTS AND LOCATIONS:
Overall Officials: Xi Wu, Principal Investigator — Huazhong University of Science and Technology
Locations (1):
- Wuhan Union Hospital, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wu X, Yang L. Quadratus Lumborum and modified Erector Spinae Plane (QLESP) block: A single-puncture technique for total hip arthroplasty. J Clin Anesth. 2020 May;61:109643. doi: 10.1016/j.jclinane.2019.109643. Epub 2019 Oct 23. No abstract available. PMID 31668470